CLINICAL TRIAL: NCT06843304
Title: The Intelligent Prevention And Control System And Strategy For The Whole Disease Cycle Of Diabetic Nephropathy
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiangmei Chen, Academician/Principal Investigator/ Clinical Professor/Director, Chinese PLA General Hospital
Other Study IDs: S2023-509-01
Record Dates: First submitted 2025-02-20; First posted 2025-02-24 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Nephropathy; T2DM
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, kidney tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes mellitus and type 2 diabetes mellitus with CKD: Based on the national multi-center diabetic nephropathy cohort built since 2017, and continues to establish prospective diabetes nephropathy whole life cycle cohort.
  Individuals with type 2 diabetes will be followed up until renal dysfunction occurs and continue to be followed up until the occurrence of renal endpoints.
  Individuals with diabetic nephropathy of type 2 diabetes will be followed up until the occurrence of renal endpoints.

SUMMARY:
Diabetic nephropathy is one of the most severe microvascular complications of diabetes and a major cause of premature death and disability. It has become a leading cause of end-stage renal failure both in China and worldwide, consuming substantial medical resources. The establishment of a comprehensive regulatory system for the development and progression of diabetic nephropathy is a critical need for effective prevention and control. However, there is a lack of representative cohorts covering the entire disease cycle of diabetic nephropathy both domestically and internationally, creating technical bottlenecks in comprehensively describing its developmental patterns. This project aims to expand and integrate existing large-sample natural population cohorts and prospective follow-up cohorts covering the entire disease cycle of diabetes and diabetic nephropathy. It will construct a panoramic life database to identify risk factors, clinical phenotypes, and multimodal biomarkers at different disease stages. By integrating multi-organ interactions (e.g., kidney, eye), the project will establish novel imaging and functional assessment technologies for microvascular complications. Utilizing artificial intelligence to process multimodal medical data, it will build and validate risk prediction models and evaluation systems for the entire disease cycle of diabetic nephropathy. The project will develop effective intelligent prevention and treatment strategies for diabetic nephropathy, promote the adoption of new technologies, and establish a medical quality control system to provide services for medical institutions. Ultimately, it aims to improve and sustain medical quality, reducing the incidence of end-stage renal disease.

ELIGIBILITY:
T2DM

Inclusion Criteria:

* Age ≥18 years old, gender is not limited
* Diagnosed with type 2 diabetes
* A history of type 2 diabetes for more than 5 years
* Negative proteinuria
* Creatinine is normal
* Good compliance, voluntarily sign informed consent

Exclusion Criteria:

* Incomplete medical records
* Lack of fundus microvascular examination or new imaging technology examination results data
* Combined with autoimmune diseases and tumors

Type 2 diabetes patients undergoing renal biopsy

Inclusion Criteria:

* Age ≥18 years old, gender is not limited
* Diagnosed with type 2 diabetes
* Kidney damage (microalbuminuria or dominant albuminuria or renal insufficiency)
* Have undergone renal puncture biopsy and have complete renal pathological diagnosis data
* Sign informed consent voluntarily

Exclusion Criteria:

* Gestational diabetes mellitus, special type diabetes mellitus
* Patients with hereditary kidney disease
* Combined with autoimmune diseases
* Diabetic nephropathy The indicators in the comprehensive assessment model of the risk of renal progression could not be obtained
* There were pregnancy plans in the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus and type 2 diabetes mellitus with CKD
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of complex renal endpoints | 3 years
  The incidence of complex renal endpoints includes eGFR decreased progressively by more than 30% from baseline, ESRD and all-cause death.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China